CLINICAL TRIAL: NCT06387875
Title: Prevention and Control of Chronic Noncommunicable Diseases in Natural Population in Qianwan New District, Ningbo
Brief Title: Cohort in Qianwan New District, Ningbo
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Ningbo Hangzhou Bay Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Hangzhou Bay Cohort
Record Dates: First submitted 2024-04-18; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Stroke; Non-Communicable Chronic Diseases
Keywords: cohort; natural population; Non-communicable Chronic Disease
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5-10ml of blood, 20ml of urine and 5g of feces were collected (if necessary) according to the chronic non-communicable disease spectrum and clinical testing needs of Qianwan New District of Ningbo; The blood samples and urine were tested for biochemistry, liver and kidney function, blood lipids and electrolytes according to clinical testing requirements, as well as multi-omics indicators as needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective is to carry out research on prevention and control of noncommunicable chronic diseases, and establish a risk prediction mechanism for chronic diseases to promote early detection, early diagnosis and early treatment of chronic diseases in natural population in Qianwan District of Ningbo, significantly reduce medical costs and extend population life span.

DETAILED DESCRIPTION:
1. Through baseline survey (cross-sectional survey) and prospective cohort design, the health status information and biological samples of residents in Hangzhou Bay Hospital were collected, and the physical, psychological and social adaptability information was collected through questionnaires and other forms, basic tests and omics measurements were carried out based on the collected samples to build a multi-dimensional data platform.
2. Develop a disease risk prediction model based on big data platform, conduct high-risk population screening and establish risk assessment files; In view of the common health problems in the study population, the key factors and effects of health status were analyzed comprehensively, and the corresponding mathematical model was established to form the prediction of health status. Finally to establish the stratified standard of population health status and provide effective health guidance.

   Questionnaire survey on epidemiology: The Hangzhou Bay Natural Population Cohort Questionnaire was designed according to the principles and requirements of cohort study. All respondents who entered the cohort will sign informed consent, receive face-to-face interview with uniformly trained investigators, and the questionnaire will be reviewed by quality control personnel for quality control.

   Physical examination: The examination contents include height, weight, blood pressure, waist circumference, hip circumference, hearing, vision, medical history and surgery, inbody composition, chest film, electrocardiogram, B-ultrasound, non-invasive arteriosclerosis examination, vascular endothelial ultrasound and other imaging examinations.

   Clinical biochemical test: 5-10 ml of blood, 20 ml of urine and 5 g of feces were collected (if necessary) according to the chronic non-communicable disease spectrum and clinical test requirements in Qianwan New District of Ningbo; The blood samples and urine were tested for biochemistry, liver and kidney function, blood lipids and electrolytes according to clinical testing requirements, as well as multi-omics indicators as needed.
3. Prospective study data: Follow-up of the cohort population (disease occurrence, death, migration, etc.) was conducted through annual active follow-up (telephone, interview, etc.) and passive follow-up, including data of all-cause death, incidence of any kind of diseases.

ELIGIBILITY:
Inclusion Criteria:

* 1) Local permanent residents aged 18 and above (including residents with household registration, or residents without household registration but with a permanent job);
* 2) No serious physical disability, can communicate normally;
* 3) Participate voluntarily and sign informed consent.

Exclusion Criteria:

* 1) Temporary resident and floating population;
* 2) There are serious health conditions unable to participate in the survey;
* 3) Those who are unwilling to accept the follow-up inspection of the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Relying on the manufacturing factories gathered around Hangzhou Bay Hospital, a relatively stable cohort of participants was provided. According to the entry criteria, eligible subjects were selected to be included in the Hangzhou Bay natural population cohort.
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
death | 4 years
  Mortality of all-cause disease were calculated by age, gender and area compared by different health management mode.
incidence of cardio-cerebrovascular diseases | 4 years
  Incidence of Cardiovascular and Cerebrovascular diseases were calculated by age, gender and area compared by different health management mode.
incidence of other non-communicable chronic diseases | 4 years
  Incidence of other non-communicable chronic diseases were calculated by age, gender and area compared by different health management mode.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD, PhD, Principal Investigator — Ningbo Hangzhou Bay Hospital
Locations (1):
- Ren Ji Hospital Afflited to School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided